CLINICAL TRIAL: NCT03791749
Title: A Randomised Controlled Trial Testing the Use of a Simple Intervention on Maternal Psychological State, Breast Milk Composition and Volume, and Infant Behaviour and Growth.
Brief Title: Mother and Late Preterm Lactation Study
Acronym: MAPLeS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS: 252031
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2020-12

CONDITIONS: Breastfeeding; Postnatal Depression; Stress, Psychological; Preterm Infant
Keywords: breastfeeding; postnatal mental health; breastfeeding support; stress; late preterm infant; breast milk
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum; Stress, Psychological; Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Support (Experimental): Home visits will be conducted at 2-3 and 6-8 weeks post-delivery. Mothers will be asked to perform a simple technique while breastfeeding at least once a day.
  Interventions: Other: Breastfeeding Support
- Standard Care (No Intervention): Home visits will be conducted at 2-3 and 6-8 weeks post-delivery. No intervention will be administered.

INTERVENTIONS:
Other: Breastfeeding Support — 12-minute simple technique
  Arms: Breastfeeding Support

SUMMARY:
Breastfeeding has various benefits for the mother and infant. It has the capability of reducing the risk of short term and long term problems for the infant, such as gastroenteritis, respiratory infections, type II diabetes and obesity, and of providing benefits for neurodevelopment. Breast milk offers even greater benefits for preterm infants. Some of the advantages of breastfeeding are related to the constituents of breast milk such as the macronutrients and bioactive factors, the hormones associated with breastfeeding such as oxytocin, and the behavioural aspects of breastfeeding (maternal sensitivity to infant cues). Despite these advantages, breastfeeding rates are below target levels mainly due to the challenges that women face that hinder breastfeeding success. Interventions aimed at improving policies, practices, and maternal support have been developed. However, other interventions that target specific modifiable barriers to breastfeeding can be useful.

The aim of this study is to investigate a simple support intervention for breastfeeding mothers of late preterm and early term infants on maternal stress reduction and infant weight gain. The investigators also aim to study the potential mechanisms by which this effect could be achieved (breast milk composition and volume, mother and infant behaviour).

ELIGIBILITY:
Inclusion Criteria:

* Mothers of late preterm infants (34 to <37 weeks) or early term infants (37 to 38 weeks)
* Intending to breastfeed for at least 6 weeks
* Free from serious illness
* Fluent in English

Exclusion Criteria:

* Currently smoking or intending to smoke while breastfeeding
* Not based in London
* Prior breast surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Maternal stress change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Stress will be measured using the Perceived Stress Scale (0 to 40 points), where higher scores indicate a higher level of perceived stress.
Infant weight change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Infant weight (kg) will be measured using an infant weighing scale.

SECONDARY OUTCOMES:
Breast milk composition (macronutrients) change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Breast milk samples will be collected at 2 and 6 weeks post-delivery. Fat, protein and carbohydrate content of breast milk (g/100 ml) will be analysed using the Miris- Human Milk Analyser.
Breast milk hormones change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Breast milk samples will be collected at 2 and 6 weeks post-delivery. Ghrelin, leptin, adiponectin and cortisol will be analysed (ng/ml) using the respective ELISA kits.
Breast milk volume change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Breast milk volume (ml) will be assessed using 48-hour test weighing
Infant behaviour change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Time spent crying and sleeping (minutes) will be measured using a 3-day behaviour diary
Infant appetite change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  Infant appetite will be assessed using the Baby Eating Behaviour Questionnaire, with the following subscales (appetite traits): General Appetite (1 to 5 points), Enjoyment of Food (1 to 5 points), Satiety Responsiveness (1 to 5 points), Food Responsiveness (1 to 5 points), and Slowness in Eating (1 to 5 points). Higher scores on each subscale indicates a greater degree of the appetite trait.
Mother-infant attachment change at 6 weeks from 2 weeks post-delivery. | Home visit 1 (2 weeks postnatally) and Home visit 2 (6 weeks postnatally)
  The extent of bonding between the mother and infant will be assessed using the Maternal Attachment Inventory (0-78 points)
Exclusive Breastfeeding Status | 6 weeks, 3 months and 6 months postnatally
  Participants will be asked whether they are still exclusively breastfeeding their infants at 6 weeks, 3 months and 6 months postnatally to assess breastfeeding status.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dib S, Wells JCK, Fewtrell M. Mother And late Preterm Lactation Study (MAPLeS): a randomised controlled trial testing the use of a breastfeeding meditation by mothers of late preterm infants on maternal psychological state, breast milk composition and volume, and infant behaviour and growth. Trials. 2020 Apr 7;21(1):318. doi: 10.1186/s13063-020-4225-3. PMID 32264947